CLINICAL TRIAL: NCT06507683
Title: A Multicenter, Single-arm, Prospective Study to Evaluate the Efficacy and Safety of Radiotherapy Combined With Ripretinib in the Treatment of Unresectable Advanced GIST
Brief Title: Evaluate the Efficacy and Safety of Radiotherapy Combined With Ripretinib in the Treatment of Unresectable Advanced GIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Zhang, Chief physician, First Affiliated Hospital of Chongqing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.0 /2024.05.01
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — ripretinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy combined with ripretinib group (Experimental): Radiotherapy (50-70Gy/25-30f)+ ripretinib(150mg QD)
  Interventions: Radiation: simultaneous integrated boost intensity-modulated radiation therapy combined with ripretinib

INTERVENTIONS:
Radiation: simultaneous integrated boost intensity-modulated radiation therapy combined with ripretinib — A cumulative radiation dose of 50 to 70 Gy is administered in 25-30 fractions, 5 fractions per week, to the target lesion(s).
  ripretinib: oral 150mg QD

SUMMARY:
The goal of this prospective study is to learn whether there is a synergistic effect when radiotherapy is combined with ripretinib in the treatment of patients with unresectable advanced GIST. It will also learn about the safety of this regimen.The main questions it aim to answer is: Dose radiotherapy combined with ripretinib prolong the time to disease progression for patients with advanced GIST?

DETAILED DESCRIPTION:
ripretinib is the standard fourth-line treatment agent for inoperable advanced GIST patients, but the mPFS is only 6.3 months. Prolonging the time to TKI resistance by using a new treatment approach is important to increase the chances of surgery ,improve the survival time, and quality of life for patients. GIST was previously thought to be a tumor that was insensitive to radiotherapy, but a growing number of studies have shown that GIST is moderately sensitive to radiotherapy and that radiotherapy is effective in controlling the tumor. In our previous work, palliative radiotherapy was given to patients with advanced GIST after multiline drug resistance, and we achieved local control for nearly 2 years while significantly improving the patient's symptoms .

In recent years, radiotherapy technology has been continuously improved, and new radiotherapy techniques can be more precise and have less impact on surrounding organs, making it possible to increase the dose of radiotherapy. For large GIST, our research team has optimized the radiotherapy technique by using simultaneous integrated boost intensity-modulated radiotherapy technique, which can deliver a safe dose at the edge of the tumor while delivering a high dose of radiotherapy at the center of the tumor, ensuring safety and resulting in better therapeutic effects.

We proposed to select some patients with unresectable advanced GIST to explore the feasibility of radiotherapy combined with TKI for the treatment of advanced GIST after failure of first-, second-, and third-line drug therapies with simultaneous addition of radiotherapy to oral ripretinib treatment

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and signed informed consent;
* age: 18 to 75 years, Male or female
* Patients with histologically confirmed GIST and Imaging evaluated as unresectable recurrent and metastatic disease or locally advanced.
* ECOG Performance Score: 0-2
* Subjects who have progressed or documented intolerance after previous first-line, second-line, and third-line treatments.
* At least one measurable lesion in the abdominal or pelvic cavity that has progressed after frontline treatment
* Adequate organ function and bone marrow reserve

Exclusion Criteria:

* estimated life-expectancy less than 3 months.
* Patients who have received previous radiotherapy to the proposed radiotherapy site, or the tumor has significant mobility, poor tolerance of radiotherapy in adjacent organs, and who are considered unsuitable for radiotherapy after MDT discussion
* Any other clinically significant comorbidities, which in the judgment of the investigator, could compromise compliance with the protocol, interfere with interpretation of the study results, or predispose the patient to safety risks.
* If female, the patient is pregnant or lactating, or plans to become pregnant during the study treatment period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Time to disease progression of irradiated lesions | Approximately 12 months since the first subject enrolled
  Time from start of radiotherapy to progression of irradiated lesions

SECONDARY OUTCOMES:
Time to disease progression of any lesions | Approximately 12 months since the first subject enrolled
  Time from start of radiotherapy to progression of any lesions
Overall survival (OS) | Approximately 12 months since the first subject enrolled
  the time from start of radiotherapy to all-cause death.
Objective Response Rate(ORR) of irradiated lesions | Approximately 12 months since the first subject enrolled
  the percentage of patients whose efficacy is confirmed as complete response(CR) or partial responses(PR) based on mRECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hayashi Y, Nguyen VTT. A narrative review of imatinib-resistant gastrointestinal stromal tumors. Gastrointest Stromal Tumor. 2021 Oct;4:6. doi: 10.21037/gist-21-10. Epub 2021 Oct 30. PMID 35814621
- [Background] Blay JY, Serrano C, Heinrich MC, Zalcberg J, Bauer S, Gelderblom H, Schoffski P, Jones RL, Attia S, D'Amato G, Chi P, Reichardt P, Meade J, Shi K, Ruiz-Soto R, George S, von Mehren M. Ripretinib in patients with advanced gastrointestinal stromal tumours (INVICTUS): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2020 Jul;21(7):923-934. doi: 10.1016/S1470-2045(20)30168-6. Epub 2020 Jun 5. PMID 32511981
- [Background] Joensuu H, Eriksson M, Collan J, Balk MH, Leyvraz S, Montemurro M. Radiotherapy for GIST progressing during or after tyrosine kinase inhibitor therapy: A prospective study. Radiother Oncol. 2015 Aug;116(2):233-8. doi: 10.1016/j.radonc.2015.07.025. Epub 2015 Jul 27. PMID 26228971
- [Background] Gatto L, Nannini M, Saponara M, Di Scioscio V, Beltramo G, Frezza GP, Ercolani G, Pinna AD, Astolfi A, Urbini M, Brandi G, Biasco G, Pantaleo MA. Radiotherapy in the management of gist: state of the art and new potential scenarios. Clin Sarcoma Res. 2017 Jan 10;7:1. doi: 10.1186/s13569-016-0065-z. eCollection 2017. PMID 28078078
- [Background] Li L, Yi X, Cui H, Zhao X, Dang J, Jiang Q, Li Y. Simultaneous Integrated Boost Intensity-Modulated Radiotherapy for Locally Advanced Drug-Resistant Gastrointestinal Stromal Tumors: A Feasibility Study. Front Oncol. 2020 Nov 23;10:545892. doi: 10.3389/fonc.2020.545892. eCollection 2020. PMID 33330024
- [Background] Cui H, Li Y, Huang W, Lu W, Yi X. Escalation of radiotherapy dose in large locally advanced drug-resistant gastrointestinal stromal tumors by multi-shell simultaneous integrated boost intensity-modulated technique: a feasibility study. Radiat Oncol. 2022 Dec 28;17(1):216. doi: 10.1186/s13014-022-02179-z. PMID 36578008
- [Background] Boruban C, Sencan O, Akmansu M, Atik ET, Ozbek S. Metastatic gastrointestinal stromal tumor with long-term response after treatment with concomitant radiotherapy and imatinib mesylate. Anticancer Drugs. 2007 Sep;18(8):969-72. doi: 10.1097/CAD.0b013e3280e94982. PMID 17667604